CLINICAL TRIAL: NCT01773213
Title: Is the Detrusor Contraction During the Ice-water-test Provoked by the Ice Water or the Rapid Bladder Filling? A Randomized, Double-blind Clinical Trial
Brief Title: Detrusor Contraction During the Ice-water-test
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Balgrist University Hospital (Other)
Responsible Party: Principal Investigator, Thomas Kessler, executive physician, Balgrist University Hospital
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 2012-0400
Record Dates: First submitted 2013-01-14; First posted 2013-01-23 (Estimated); Last update posted 2018-03-05 (Actual); Status verified 2018-03

CONDITIONS: Urinary Bladder, Neurogenic; Neuropathic Bladder
Keywords: Lower urinary tract; Bladder; Neuropathic bladder; Overactive bladder
MeSH Terms: conditions — Urinary Bladder, Neurogenic; Urinary Bladder, Overactive

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Bladder dysfunction, ice-water-test (Other)
  Interventions: Procedure: Ice-water-test
- Bladder dysfunction, warm water-test (Other)
  Interventions: Procedure: Ice-water-test

INTERVENTIONS:
Procedure: Ice-water-test

SUMMARY:
In this randomized, double-blind clinical trial including patients with a neurogenic lower urinary tract dysfunction undergoing urodynamic investigation at the Spinal Cord Injury Center, Balgrist University Hospital, Zürich, we aim to investigate whether the detrusor contraction during the ice-water-test is provoked by the ice water or the rapid filling.

DETAILED DESCRIPTION:
The ice-water-test (IWT) was first described 1957 by Bors and Blinn and it was thought to differentiate between lesions of the upper and lower motoneuron. In cat studies, it was shown that the IWT is a C-fiber mediated lower motoneuron segmental reflex and that these unmyelinated C fibers are associated with cold receptors. This explains the positive IWT in patients with upper motoneuron lesions. In healthy humans, the IWT is positive up to the age of 4 years and becomes negative thereafter since the reflex is centrally inhibited. However, this reflex might be unmasked by a neurological disease and/or injury.

Considering that C-fibers are involved in the pathogenesis of detrusor overactivity, the IWT seems to be a useful diagnostic tool in daily practice. However, although there are many studies published on the IWT, it is unclear whether the detrusor contraction during the IWT is provoked by the ice water or whether it might be caused by the rapid filling. Therefore, we designed this randomized, double-blind trial.

ELIGIBILITY:
Inclusion Criteria:

* neurogenic lower urinary tract dysfunction
* urodynamic investigation
* written informed consent
* ≥ 18 years old

Exclusion Criteria:

* symptomatic urinary tract infection
* < 18 years old
* ≥ 90 years old
* no written informed consent
* pregnancy

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2012-12; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Increase of detrusor pressure in cmH20 | 60 minutes
  Increase of detrusor pressure during the verum ice-water-test and the placebo ice-water-test (intravesical pressure increase during the filling of the bladder with 4°C or 36°C water)

SECONDARY OUTCOMES:
Sensations (yes/no) | 60 minutes
  Coldness, Urgency, Pain, Information with yes or no
Urinary incontinence | 60 minutes
  Urinary incontinence during the test
Heart rate | 60 minutes
  Assessment of the heart rate during the test

CONTACTS AND LOCATIONS:
Locations (1):
- Neuro-Urology, Spinal Cord Injury Center & Research, Balgrist University Hospital, Zurich, Switzerland